CLINICAL TRIAL: NCT03937232
Title: Mirrored Movement Compared to Cross-education for Recovery After Hand or Wrist Injury: a Pilot Study.
Brief Title: Mirrored Movement Compared to Cross-education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Tara Packham, Assistant Professor, McMaster University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 5979
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Hand Injuries
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Intervention Model Description: Cross-education OR Mirror visual feedback OR Cross-education + mirror visual feedback OR usual care
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cross-Education (Active Comparator): Cross education has been defined as the unilateral training of a limb with resisted exercise for the benefit of transferring strength to the contralateral (often injured or immobilized) limb. Participants randomized to cross-education will be provided with a hand-grip strengthener, adjusted to provide resistance at 70-80% of their maximum grip strength. They will be given written, illustrated instructions for performing grip strengthening exercises for their uninjured hand in a seated position with both forearms comfortably supported; this will be demonstrated during the teaching session. The instructions will ask for the participant to complete 3 sets of 10 repetitions twice daily, with additional instructions for appropriate grading of resistance. A diary for tracking exercise completion and attendance for usual care will also be provided.
  Interventions: Behavioral: Cross-Education; Other: Usual care
- Mirror Visual Feedback (Active Comparator): Mirror visual feedback is the performance of movements with an uninjured hand in front of a mirror hiding the injured hand, thus creating the illusion of bilateral movement. Participants randomized to mirror visual feedback will be provided with a portable mirror and stand, and instructed with accompanying demonstration on how to set up on a table for comfortable visualization. They will be given written, illustrated instructions for performing mirror visualization of exercises completed by the uninjured hand only from a position of neutral rotation of the forearm. The instructions will ask for the participant to complete a three sets of 10 repetitions for finger flexion and extension (mimicking the fisting motion of the grip strengthening exercises) twice daily. A diary for tracking exercise completion and attendance for usual care will also be provided.
  Interventions: Behavioral: Mirror Visual Feedback; Other: Usual care
- Cross-education + Mirror Visual Feedback (Experimental): In this group, participants will perform the cross-education resistance exercise in front of the mirror, visualizing the performance of the resistance exercises. Participants randomized to cross education with mirror visual feedback will be provided with both a hand-grip strengthener and a portable mirror and stand, and instructed with accompanying demonstration on how to set up on a table for comfortable visualization. They will be given written, illustrated instructions for performing mirror visualization hand grip strengthening exercises completed by the uninjured hand only from a position of neutral rotation of the forearm. The instructions will ask for the participant to complete 3 sets of 10 repetitions twice daily, with additional instructions for appropriate grading of resistance. A diary for tracking exercise completion and attendance for usual care will also be provided.
  Interventions: Behavioral: Mirror Visual Feedback; Other: Usual care
- Usual Care (Active Comparator): Participants randomized to usual care will be encouraged to attend the recommended rehabilitation, and provided with a diary for frequency of rehab attendance, and tracking any exercises completed at home.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Cross-Education — Home exercise program + usual care
  Arms: Cross-Education
Behavioral: Mirror Visual Feedback — Home exercise program + usual care
  Arms: Cross-education + Mirror Visual Feedback; Mirror Visual Feedback
Other: Usual care — Hand rehabilitation provided by occupational therapists and physiotherapists in a multidisciplinary outpatient setting

SUMMARY:
Recovery after a hand or wrist injury often includes wearing a cast, or limiting daily activities to help with healing, but this may lead to deconditioning. Previous research suggests resistance training with the healthy arm during this period could help improve recovery of the injured arm: this is called cross-education. Mirror visual feedback (e.g. watching the movement of an uninjured hand in front of a mirror hiding the injured hand to create the illusion both hands are moving) is another cross-body method which can improve recovery after stroke, and prevent or reduce pain in complex regional pain syndrome. Both of these treatments may work because they activate a specific area in the brain: using them together might strengthen the effects. However, this has never been studied after injury. The investigators are proposing a pilot study to see if it is possible and helpful to use these treatments in combination to improve recovery of grip strength and reduction of pain and disability. The investigators will use this information as a foundation to tell us how to run the best study to test these ideas in ways to be confident in the results.

DETAILED DESCRIPTION:
When someone has an injury to the hand or wrist, often the person's doctor and therapists will ask them to use a cast or a splint to protect the body while it heals. They also may ask the person not to do certain movements, or any activities where it is necessary to use the hand for squeezing or gripping. This is important to allow healing, but the injured arm can become weaker during this period. New research has demonstrated that performing specific forms of exercise on the uninjured side can help speed recovery on the injured side, even when the injured hand is still in a cast.

Two of these types of exercise are called cross-education and mirror visual feedback. Cross-education means doing resistance or strengthening exercises on the uninjured side while the injured side is resting. Mirror visual feedback is performing exercise or movements with the uninjured hand in front of a mirror, hiding the injured hand resting behind the mirror, so it looks like the injured hand is doing the exercises too. The investigators think both of these exercises work because they use the same part of the brain, part of our movement control network that helps us coordinate movements on both sides of the body. Perhaps they might work even better if used together.

This study will test cross-education, mirror visual feedback or cross-education combined with mirror visual feedback added to the usual therapy after a hand or wrist injury. The investigators need to be sure that this is better than usual care, so some people who participate in the study will just have the usual care, and not do any extra exercise. Because limited research has been done on these methods after injury, this will be a small study to test the best ways to run a big study that will provide solid proof about these ideas. That means the investigators will ask participants to keep track of how often they do their exercises, and to tell the study team about any problems or concerns they have when they are doing their exercises.

If it can be demonstrated that cross-exercise and/or mirror visual feedback can speed up or improve recovery after a hand or wrist injury, it might help participants get back to work and their usual activities faster and with less pain. These treatments don't cost a lot of money or need a lot of special equipment, so they could be used in many different countries. If the study can show these exercises help with hand and wrist injuries, they might also be able to be used for therapy after stroke, or with other kinds of injuries like foot and ankle fractures.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or older
* Acute injury to one hand or wrist requiring protection or immobilization, including fractures (managed conservatively or with surgery), tendon laceration/repairs, burns, and/or ligament injuries/repairs
* Able to provide informed consent

Exclusion Criteria:

* Unable to complete study questionnaires in English
* Traumatic injuries to other limbs or axial skeleton (e.g. whiplash, rib fracture, concurrent lower limb injury)
* Anticipates difficulty to return for follow-up visits (i.e. out of catchment)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Trial feasibility | 3 months
  total number of potential participants vs. enrolled participants from the clinic

SECONDARY OUTCOMES:
Composite finger flexion | 1, 2, and 3 months
  the distance (in cm) from the junction of the nail fold on the fingertip to the distal palmar crease on the hand for the index, middle, ring and small fingers
Patient-Rated Wrist and Hand Evaluation | 1,2,and 3 months
  This patient self report measure is scored from 0-100 across two subscales containing 15 items addressing pain and disability in the hand and wrist. Higher scores indicate more pain and disability.
Pain Catastrophizing Scale | 3 months
  This patient self-report measure contains 14 items addressing negative pain beliefs. It is scored from 0-52, with a score of over 30 considered to represent unhelpful beliefs about pain.
Hand grip strength | 3 months
  Grip strength as measured by hand dynamometer (in kilos).
Adverse events | 3 months
  Number of major adverse events defined as need for secondary surgical intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green LA, Gabriel DA. The cross education of strength and skill following unilateral strength training in the upper and lower limbs. J Neurophysiol. 2018 Aug 1;120(2):468-479. doi: 10.1152/jn.00116.2018. Epub 2018 Apr 18. PMID 29668382